CLINICAL TRIAL: NCT00778440
Title: Risk Level of Suffering From Traffic Injury in Primary Health Care: LESIONAT Project
Acronym: LESIONAT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Unitat de Suport a la Recerca, Barcelona, Spain (Other); Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other)
Responsible Party: Dr Carlos Martin, Unitat Suport Recerca Àmbit Atenció Primària Barcelona Institut Catala Salut
Other Study IDs: PI08/90242
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Traffic Accident; Chronic Disease; Prevalence of Psychoactive Substances in Road Traffic; Relative Risk Estimation of Accident for Impaired Drivers
Keywords: Injuries; Traffic Injuries; Preventive medicine; Observational studies; Primary care
MeSH Terms: conditions — Chronic Disease; Wounds and Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Main objectives:

* To know the distribution of risk elements of traffic injuries

Secondary objectives:

* To study the distribution of risk elements related with the possibility of suffering from a TI in relation to medication, chronic health problems, and consumption of psychoactive substances (alcohol and others).
* To know the relation between levels of perception of risk of suffering from a TI and the presence of chronic problems, medications, or consumption of psychoactive substances.

DETAILED DESCRIPTION:
Methodology:

Design: Observational, transversal, and multicentric research

Field of study: 20 PHC users from urban areas

Population of study: random consecutive sampling of ≥ 16 years old drivers with open medical history.

Measure's tools: Two means for data collection: survey among health professionals with medical history and structured telephonic survey about behaviours and risk perceptions in drivers.

Variables: Sociodemographic data, chronic pathologies related to TI, consumption of medications ,Alcohol consumption (AUDIT-C test), Psychoactive substances consumption (self declared), Level of perception of risk according to professionals.

Telephone survey: Class and age of driving license, Type of roads, Weekly driving time, Safety behaviours, Record of collisions/injuries in last year,Self perception of health level(SF-12) andSelf perception of risk level.

An descriptive analysis of population will be performed, a distribution of risk elements associated to TI will be described through bivariant analyses, and for describing the factors associated to perceived risk levels a linear regression multiple model will be built.

ELIGIBILITY:
Inclusion Criteria:

* 16 years old or more
* Catalan and/or spanish language speakers
* Drivers with driver license
* Participation accepted by the patient

Exclusion Criteria:

* Patients who do not have contact phone number.
* Patients who do not answer up to 3 phone calls
* Patients with severe mental or physical health disorder

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: drivers with active medical records of 16 years old or more
Sampling Method: Probability Sample
Enrollment: 1540 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Martin, MD, PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- Unitat Suport Recerca Barcelona. IDIAP Jordi Go, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Martin-Cantera C, Prieto-Alhambra D, Roig L, Valiente S, Perez K, Garcia-Ortiz L, Bel J, Marques F, Mundet X, Bonafont X, Birules M, Soldevila N, Briones E; LESIONAT Research Group. Risk levels for suffering a traffic injury in primary health care. The LESIONAT project. BMC Public Health. 2010 Mar 16;10:136. doi: 10.1186/1471-2458-10-136. PMID 20233403